CLINICAL TRIAL: NCT02115009
Title: Comparative Study of The Relationship Between the Sacroiliac Joint (SIJ) and Lumbopelvic Configurations With SIJ Nerve Entrapments and Chronic Low Back Pain
Brief Title: The Sacroiliac Joint With SIJ Nerve Entrapments and Chronic Low Back Pain
Acronym: SARA31143
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Natan Peled, Prof. Nathan Peled, Carmel Medical Center
Other Study IDs: CMC-13-0072-CTIL
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Low Back Pain
Keywords: sacroiliac joint lumbopelvic ,chronic low back pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall goal of this study is to characterize the SIJ form, function, nerve entrapments, lumbo-pelvic configuration and their possible relationships with nonspecific chronic LBP in females and males. Specific aims: 1.To investigate the relationship between SIJ bridging and NSCLBP in females and males. 2. To investigate the prevalence and characterization of nerve entrapment of the lumbar sacral plexus around the SIJ in females and males. 3. To investigate the correlation between the lumbar sacral plexus nerve entrapments around the SIJ and NSCLBP in females and males. 4. To investigate the relationship between the lumbar sacral plexus nerve entrapments around the SIJ and lumbo-pelvic morphology in females and males. 5. To characterize the location and severity of articular degenerative changes in the SIJ and its relationship with lumbo-pelvic morphology in females and males. 6. To investigate the relationship between articular degenerative changes in the SIJ and LBP in females and males.

DETAILED DESCRIPTION:
Background: Low back pain is a major cause of disability among the working population significantly impacting the socioeconomic status. Pelvic girdle structures, mainly the sacroiliac joint, may act as major factors in LBP. The interaction, however, between possible adjacent nerve entrapments around the SIJ, osteological changes in the SIJ and their relationship with the lumbo-pelvic configuration in patients with and without nonspecific chronic LBP is still unclear. Studying this interaction radiologically, histologically, anatomically and clinically will significantly improve our understanding of the pathophysiology of lumbo-pelvic pain and improve its diagnosis and medical treatment.

Methods: The research project includes four major studies: Radiological and clinical studies- Computerized tomography images of the lumbo-pelvic region of 200 individuals age range 20-50 years, admitted to the Carmel Medical Center with and without LBP will be examined prospectively to evaluate the relationship between the SIJ structures, lumbo-pelvic nerve pathways, lumbo-pelvic configuration and SIJ osteological changes. The presence and prevalence of nerve entrapments in these phenomena will be assessed using a CT software distance measurement tool. All individuals will be referred by their physicians for CT regardless the purposes of the current study thus no extra radiations will be required. Inclusion criteria for the NSCLBP group are individuals with pain in the lower back region, pelvic area, hips, groin, abdominal, buttocks, and thighs. Individuals with the following spinal conditions will be excluded: Any level of lumbar disc bulging, spondyloarthropathy, diffuse idiopathic skeletal hyperostosis, spinal tumors, osteoporotic fractures, traumatic vertebral fractures, and previous spinal surgeries. All CT images will be obtained from the Department of Radiology, and will be analyzed at the Spinal Research Lab. The interaction between the above mentioned radiological parameters and clinical self-reported lumbo-pelvic pain questionnaires will be assessed. Anatomical/histological studies - The morphological study of the lumbo-pelvic nerve pathways will be carried out on human cadavers at the Tel-Aviv University. The histological study of the SIJ microstructure will be carried out on samples taken from human cadavers at the Department of Anatomy, TAU.

ELIGIBILITY:
Inclusion Criteria:

-For the NSCLBP group - subjects with pain in the lower back region, pelvic area, hips, groin, abdominal, buttocks, and thighs

Exclusion Criteria:

-Subjects with any level of lumbar disc bulging, spondyloarthropathy, diffuse idiopathic skeletal hyperostosis, spinal tumors, osteoporotic fractures, traumatic vertebral fractures, and previous spinal surgeries

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects (100 males and 100 females) with and without Low Back Pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of the recruited participants | 1 year
  1 year after the starting point of the study the investigators are expecting at least 35% recruiting of the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Peled, MD, Principal Investigator — Carmel Medical Center